CLINICAL TRIAL: NCT04674293
Title: Russian Prospective Multicenter Registry Study of Intravenous Thrombolytic Therapy for Acute Ischemic Stroke.
Acronym: IVT-AIS-R
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Principal Investigator, Mikhail Soldatov, Researcher, Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health
Other Study IDs: IVT-AIS-R
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: The Aim the Study is to Collect and Analyze Data on Patients With Acute Ischemic Stroke During Intravenous Thrombolytic Therapy With Alteplase

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Revelisa — Thrombolytic therapy for patients with ischemic stroke

SUMMARY:
Russian prospective multicenter registry study of intravenous thrombolytic therapy for acute ischemic stroke.

DETAILED DESCRIPTION:
1. RATIONALE FOR THE STUDY 1.1. The urgency of the problem Cerebral stroke ranks second in the frequency of deaths from diseases of the circulatory system in the Russian Federation. Mortality rates from cerebrovascular diseases are among the highest in the world (175 per 100 thousand population) and, unlike most economically developed countries, not only do not decrease, but also tend to increase. The annual death rate from a stroke in Russia is one of the highest in the world (175 cases per 100 thousand population per year). The early 30-day mortality rate after stroke is 34.6%, and about 50% of patients die within a year, i.e. every second sick [1].

   International experience shows that a decrease in mortality from cardiovascular diseases is achieved as a result of the implementation of coordinated complexes, the main of which are raising the awareness of the population about the risk factors of vascular diseases and their prevention, the introduction of effective preventive programs and the improvement of the system of medical care in stroke. stroke include the use of modern highly effective methods of reperfusion of the brain substance in the first hours of the disease, aimed at restoring blood flow in the affected vessel, which allows to prevent the development of irreversible damage to the brain substance or to reduce its volume, i.e. to minimize the severity of residual neurological deficit [2].

   The safety and efficacy of systemic thrombolysis in ischemic stroke using rt-PA (alteplase) has been proven in a number of large randomized placebo-controlled clinical trials (NINDS, ECASS I, II, III, ATLANTIS) [3], as well as the SITS-MOST and SITS-ISTR registers [4 , 5]. According to the recommendations of the European Stroke Organization (ESO) and the American Stroke Association (ASA), systemic thrombolytic therapy (TLT) using rt-PA (alteplase) is the most effective treatment for ischemic stroke in the first 4.5 hours from the onset of the disease [6, 7].

   1.2. Rationale for the study To date, two alteplase preparations are registered in the Russian Federation - Revelisa® (JSC GENERIUM, Russia) and Actilyse® (BoehringerIngelheimPharma GmbH and CoKG, Germany). The information obtained in this register will help to clarify the data on the use of thrombolytic therapy in patients with acute ischemic stroke in the Russian Federation.
2. PURPOSE AND OBJECTIVES OF THE RESEARCH 2.1. Purpose of the study The aim of this study is to collect and analyze data on patients with acute ischemic stroke during intravenous thrombolytic therapy with alteplase (Revelisa®) in routine clinical practice.

   2.2. Research objectives
   * Collecting and analyzing data on patients with acute stroke who received TLT in routine clinical practice;
   * Obtaining data on the outcomes of AII in patients who received TLT in routine clinical practice;
   * Obtaining data on the complications of TLT in patients with acute ischemic stroke in routine clinical practice.
3. RESEARCH DESIGN This study is an open, prospective, multicenter, non-interventional (registry) study.

   This study does not provide for any interference with normal clinical practice, including the use of investigational therapy or special research methods. The physician will collect data on all patients with acute ischemic stroke who are admitted to the hospital and who meet the inclusion criteria for this study, starting from 1 July 2019.
4. SELECTION AND EXCLUSION OF RESEARCH SUBJECTS 4.1. Description of the study population The study will include all patients of any gender and age with a confirmed diagnosis of stroke of ischemic type (AII) who meet the selection criteria for the study and hospitalized in specialized hospitals. At least 500 patients are planned to be included in the study.

4.2. Inclusion criteria

To be included in the study, patients must meet the following criteria:

1. Patients of any gender and age with a confirmed diagnosis of ischemic stroke (AII);
2. Carrying out the patient with intravenous thrombolytic therapy with the drug alteplase (Revelisa®).

5. SURVEY MANAGEMENT The principal investigators of the centers are responsible for conducting research at each specific clinical center. The national project coordinator is prof. Shamalov N.A. Operational project management and statistical analysis is carried out by Generium JSC, database maintenance and data management will be carried out on the basis of the ROSMED.INFO online medical platform, medical monitoring will be carried out by the Federal Center for Cerebrovascular Pathology and Stroke of the Ministry of Health of the Russian Federation.

6. THERAPY The use of any investigational drug is not foreseen in this register. All patients included in the study will receive thrombolytic therapy with drugs registered in the Russian Federation, and in accordance with

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, patients must meet the following criteria:

1. Patients of any sex and age with a confirmed diagnosis of ischemic stroke (AII);
2. Carrying out the patient with intravenous thrombolytic therapy with the drug alteplase (Revelisa®).

   -

   Exclusion Criteria:

   -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients of any gender and age with a confirmed diagnosis of ischemic stroke (AII), who meet the selection criteria for the study and are admitted to specialized hospitals. At least 500 patients are planned to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The overall frequency of a favorable clinical outcome (from 0 to 2 points on the modified Rankin scale) [30 ± 7 days and 90 ± 7 days after TLT]; | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution "Federal Center for Brain and Neurotechnologies" of the Federal Medical and Biological Agency, Moscow, Ostrovityanova Street, 1, P. 10, Russia

IPD SHARING:
Plan to Share IPD: Undecided